CLINICAL TRIAL: NCT02877290
Title: The Effect of Non-invasive Ventilation on the Oxygenation of Peripheral Muscle Tissue, Cardiovascular System and Exercise Capacity in Hypercapnic COPD Patients
Brief Title: The Effect of Non-invasive Ventilation on the Oxygenation of Peripheral Muscle in Hypercapnic COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: ResMed (Industry)
Responsible Party: Principal Investigator, Klaus Kenn, Prof. Dr. Klaus Kenn, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NIV/NIRS in exercise
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: COPD; Hypercapnia
Keywords: COPD; NIRS; NIV; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia; Motor Activity | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cycling test first with NIV, then without NIV (Experimental): patients in this arm will perform their first constant work rate test while using NIV and the second constant work rate test without NIV
  Interventions: Device: non-invasive ventilation (NIV)
- cycling test first without NIV, then with NIV (Experimental): patients in this arm will perform their first constant work rate test without NIV and the second constant work rate test with NIV
  Interventions: Device: non-invasive ventilation (NIV)

INTERVENTIONS:
Device: non-invasive ventilation (NIV)

SUMMARY:
In this study, 20 hypercapnic COPD patients will perform two constant workrate endurance cycle tests. One test will be while using non-invasive Ventilation (NIV) support, one without in a randomized cross-over design. The aim is to measure, whether NIV is able to change peripheral and respiratory muscle oxygenation.

DETAILED DESCRIPTION:
In this study patients will perform one incremental work rate test to obtain peak work rate. On the following days two constant work rate cycle endurance tests (CWRT) will be performed at 60% of Peak work rate using a randomised cross-over design. Between the two CWRTs there will be one hour of recovery time in between.

One of the CWRTs will be performed with the support of non-invasive Ventilation (NIV), the other one without. Respiratory and cardiovascular parameters will be observed through transcutaneous measurement of CO2 (Sentec device) and near-infrared spectroscopy devices.

The purpose of this study is, to examine whether the use of NIV not only decreases patients dyspnoea, but also has positive effects on the patients cardiovascular System, exercise capacity and muscle oxygenation. The investigators will examine the tissue oxygen saturation in the 7th intercostal space (reflecting a respiratory muscle) and on the M. vastus lateralis of the leg during both CWRTs. With the Support of NIV, it is expected to see a change in the oxygenation towards a better perfusion of the leg muscle, due to a facilitation of the work of breathing. This may result in a later onset of leg fatigue and an increased exercise capacity of the patients. To have an equivalent workload all parameters will be compared during isotime.

To conclude, aim of this study is to record the interplay of Oxygenation and Perfusion between the Intercostal muscles and the peripheral leg muscle during exercise. The investigators hypothesize, that the use of NIV may change the oxygenation in favour of the leg muscle through relieving the respiratory muscles.

ELIGIBILITY:
Inclusion Criteria:

* Chronic obstructive pulmonary disease GOLD (Global initiative for chronic obstructive lung disease) stage IV
* Hypercapnia: pCO2>50mmHg (at rest or in exercise)
* written consent

Exclusion Criteria:

* orthopaedic comorbidities that do not allow a cycle endurance test
* acute exacerbation of COPD
* Cardiac insufficiency, acute coronary syndrome

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
cycle endurance time | maximum 20 minutes
  time patient ist able to cycle at 60% of his peak work rate

SECONDARY OUTCOMES:
Borg scale of dyspnoea | 30 minutes
  In the beginning and in the end of the constant work rate tests patients will be asked to rate their current level of dyspnoea on the modified Borg scale from 0 to 10
Borg scale of leg fatigue | 30 minutes
  In the beginning and in the end of the constant work rate tests patients will be asked to rate their current Level of leg fatigue on the modified Borg scale from 0 to 10
Oxygen saturation | 30 minutes
  Measurement of the oxygen saturation during the constant work rate tests
Heart rate | 30 minutes
  Measurement of the heart rate during the constant work rate tests using a pulse oximeter
Arterial blood pressure | 30 minutes
  Riva-Rocci measurement of the arterial blood pressure before and in the end of the constant work rate tests
arterial carbondioxide partial pressure | 30 minutes
  recording of the transcutaneously measured arterial carbondioxide partial pressure using Sentec technology during the constant work rate tests
Tissue Saturation Index | 30 minutes
  the near infrared technology delivers the Tissue Saturation Index throughout the constant work rate test
total hemoglobin | 30 minutes
  the near infrared technology delivers the Tissue Saturation Index throughout the constant work rate test

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Prof. Dr., Principal Investigator — Schoen Klinik BGL
Locations (1):
- Schoen Klinik BGL, Schoenau Am Königssee, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gloeckl R, Andrianopoulos V, Stegemann A, Oversohl J, Schneeberger T, Schoenheit-Kenn U, Hitzl W, Dreher M, Koczulla AR, Kenn K. High-pressure non-invasive ventilation during exercise in COPD patients with chronic hypercapnic respiratory failure: A randomized, controlled, cross-over trial. Respirology. 2019 Mar;24(3):254-261. doi: 10.1111/resp.13399. Epub 2018 Sep 21. PMID 30242790